CLINICAL TRIAL: NCT03845426
Title: Factors Affecting the Pulpal Prognosis of Injured Teeth
Acronym: TRAUMA
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC18118
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Dental Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Root canal treatment. — Once pulpal necrosis has been diagnosed, root canal treatment will be carried out by the patient's general practitioner. This is an end point for the tooth in the study.

SUMMARY:
Factors affecting the pulpal prognosis of injured teeth. Dental injuries may affect the survival of teeth. It is recommended to monitor the injured teeth at regular intervals to ensure that the appropriate treatment is delivered promptly. In order to conclude what treatment is required, a correct diagnosis must be reached.

However, reaching this diagnosis can be difficult as injured teeth often respond erroneously to many of the diagnostic tests used, thereby affecting our ability to interpret the results.

This study aims to identify the clinical factors that affect the ability of the blood supply of a tooth to survive an injury. This will help ensure that patients are provided with the appropriate treatment with the avoidance of delays that may affect the long-term survival of the tooth.

Patients that attend the Edinburgh Dental Institute trauma clinic will be invited to participate in this study. The patients, seen on this clinic, are assessed in regular intervals in a systematic way, as per accepted and validated international guidelines on the subject of dental trauma. There are specific investigations and clinical assessments that are carried out on the initial and each review appointment.

The study will attempt to identify those teeth that lose their vitality at different points following the injury and will attempt to link this to the nature of the injury suffered. The data will be collected from the patients' routine dental trauma assessment and no additional investigations will be required. As per routine practice the patients are reviewed for one year following their injury unless otherwise indicated. All responses to the investigations will be collected and combined to identify the prognostic factors associated with the loss of vitality of traumatised teeth.

DETAILED DESCRIPTION:
Dento-alveolar trauma may affect the quality of life of patients and the long term prognosis of the teeth. Following dental trauma regular monitoring and follow up of the teeth is required to ensure that the appropriate treatment is delivered promptly. Although there is information in the literature focused on child and adolescent dental trauma, there is limited information regarding traumatised permanent teeth. Permanent teeth have differing healing capacity after injury and this is dependent on the degree of root formation.

During the initial assessment of patients that have suffered from dental trauma, negative responses to investigations assessing the health of the vasculature might lead clinicians to initiate unnecessary and irreversible treatment on traumatised teeth. Equally false positive results might delay treatment which might have an effect on the outcome, leading to the development of healing complications such as infection and root resorption. By collecting and analysing the clinical factors, we aim to identify which of aspects of the assessment might influence the prognoses of the teeth.

ELIGIBILITY:
Inclusion Criteria:

* patients that have suffered dental trauma (lateral luxation)
* patients must have attended the Dental Trauma clinic within 2 weeks form the presenting injury
* patients should re-attend for review and monitor of teeth for at least 3 months following the injury
* patients older than 16 years old
* patients that have signed the informed consent

Exclusion Criteria:

* patients presented more than 2 weeks following the injury
* patients suffered from injuries other than lateral luxation
* patients younger than 16 years old
* adults with incapacity
* patient that have not consented to take part

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the dental trauma clinic, which runs every Monday in Edinburgh Dental Institute.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Pulpal necrosis | 3 months
  Number of participants developing pulpal necrosis following lateral luxations tooth injuries

CONTACTS AND LOCATIONS:
Overall Officials: Robert Philpott, BDS,, Principal Investigator — bob.philpott@ed.ac.uk
Locations (1):
- Edinburgh Dental Institute, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided